CLINICAL TRIAL: NCT06990568
Title: The Effect of Probiotic Administration on the Incidence of Antibiotic-associated Diarrhea in Patients With Community-acquired Pneumonia
Brief Title: Impact of Probiotics on Antibiotic-associated Diarrhea in Community-acquired Pneumonia
Acronym: PROBIO
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: National Health Insurance Service Ilsan Hospital (Other)
Responsible Party: Principal Investigator, Eunki Chung, MD, National Health Insurance Service Ilsan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2025-01-010; NHIMC-2024-CR-070 (Other Grant/Funding Number: National Health Insurance Service Ilsan Hospital)
Record Dates: First submitted 2025-05-16; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Pneumonia; Probiotics; Diarrhea
MeSH Terms: conditions — Pneumonia; Diarrhea

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Lacidofil (Experimental): Take 1 capsule of Lacidofil in the morning and evening after meals, for a total of 2 times a day. The total duration of the dosage is the antibiotic treatment period plus 5 days.
  Interventions: Drug: Lacidofil
- Placebo (Placebo Comparator): Take 1 capsule of placebo in the morning and evening after meals, for a total of 2 times a day. The total duration of the dosage is the antibiotic treatment period plus 5 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lacidofil — 1 capsule twice daily.
  Arms: Lacidofil
Drug: Placebo — 1 capsule twice daily.
  Arms: Placebo

SUMMARY:
The study goal is to determine whether oral administration of a probiotic mixture can reduce the incidence of antibiotic-associated diarrhea in patients with community-acquired pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 19 years or older admitted with a diagnosis of community-acquired pneumonia
* Patients eligible for oral medication administration (able to take oral or enteral feeding)

Exclusion Criteria:

* Sepsis patients
* Patients admitted to the intensive care unit (ICU) following endotracheal intubation
* Elderly patients aged 80 years or older
* Pregnant women
* Patients who have diarrhea at the time of admission
* Patients with a history of using probiotics within 3 months prior to admission
* Patients with a history of using laxatives within 1 week prior to admission
* Patients suspected of being in shock (mean arterial pressure < 65 mmHg) at the time of admission

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of antibiotic-associated diarrhea | Within 14 days after the cessation of Lacidofil or placebo administration
  Antibiotic-Associated Diarrhea (Definition: Occurrence of diarrhea more than 3 times a day, occurring at least 24 hours after the first administration of antibiotics)
  * Diarrhea is defined using the Bristol Stool Form Scale (BSF) as BSF 6 or 7. BSF 6: Mushy stool [Soft pieces with ragged edges, mushy stool] BSF 7: Watery stool [Liquid-like, no solid form, completely liquid]

SECONDARY OUTCOMES:
Occurrence of Clostridium difficile infection | Within 14 days after the cessation of Lacidofil or placebo administration
  Positive result in Clostridium difficile test: toxin, X-pert, or culture
Total length of hospitalization | Within 14 days after the cessation of Lacidofil or placebo administration
  the duration from admission to discharge
Duration of antibiotic use | Within 14 days after the cessation of Lacidofil or placebo administration
  period of antibiotic use during hospitalization + duration of oral antibiotic use after discharge

IPD SHARING:
Plan to Share IPD: No